CLINICAL TRIAL: NCT05459363
Title: Improved Training Happens With Integrated Neuromuscular and Cognitive Challenge
Brief Title: Neuromuscular Cognitive Training
Acronym: I-THINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ke'La H Porter (Other)
Responsible Party: Sponsor-Investigator, Ke'La H Porter, Research Assistant, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 76666
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Injury;Sports
Keywords: injury prevention; cognition; physical performance; postural stability; neuromuscular
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Varsity Athletes (Experimental): Healthy adults recruited from the University of Kentucky varsity tennis programs.
  Interventions: Other: I-THINC

INTERVENTIONS:
Other: I-THINC — Improved Training Happens with Integrated Neuromuscular and Cognitive Challenge (I-THINC) is an injury prevention program. It will be used to integrate cognitive tasks with traditional sports injury prevention approaches that focus on balance, agility, and neuromuscular control.

SUMMARY:
This project will utilize a quasi-experimental, multiple baseline pretest-posttest design where participants will complete postural stability assessments, physical performance assessments, and questionnaires to evaluate perceptions toward injury prevention before and after completing a 6-week neuromuscular-cognitive prevention program.

DETAILED DESCRIPTION:
The I-THINC program will address aspects of cognition (i.e., reaction time/processing speed, working memory, cognitive flexibility, inhibitory control, attention, and dual-tasking) while completing common movement patterns utilized in tennis (i.e., lateral shuffle, rapid acceleration/deceleration, and postural stability). The proposed program will take place in the participants training facility. The program will be implemented twice per week for six weeks (12 sessions) with each session lasting 20 minutes. To add variety, there will be two complementary programs (A and B) comprising of four exercises increasing in complexity every two weeks. Each week participants will complete Program A during the first session and Program B during the second session.Exercises will progressively challenge cognitive and physical demand. Exercises were designed to address the most common injuries in tennis.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults from the University of Kentucky varsity tennis programs

Exclusion Criteria:

* not medically cleared for participation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Change in single task static postural stability | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Single task static postural stability will be assessed with an Accusway Plus force plate.
Change in dual task postural stability | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Dual task static postural stability will be assessed with an Accusway Plus force plate while completeing an upper extremity reaction time on the Dynavision D2.
Change in dynamic postural control | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Dynamic postural control will be assessed with the single leg hop.
Change in dual task dynamic postural control | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Dynamic postural control will be assessed with the single leg hop. An additional cognitive task - responding to LED color cues - will be added.
Change in speed, power and agility (single measure) | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Speed, power and agility will be measured using the Run Decide Test.
Change in reactive agility | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Reactive agility will be assessed with the 4x4 box drill.
Change in lower extremity reaction time | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Lower extremity reaction time will be assessed with the lower extremity reaction test, deactivating sensors as quickly as possible with their foot.
Change in HBMS | 6 weeks (baseline, one week after baseline, and immediately following the 6 week intervention)
  Health Belief Model Scale (HBMS) is used to assess behavioral determinants of exercise related injury prevention programs and is comprised of six subscales: susceptibility, severity, benefits, barriers, cues to action, and self-efficacy. Participants rate how strongly they agree or disagree with the statements on a Likert scale ranging from 3 to -3, with a 3 indicating strongly agree and -3 indicating strongly disagree. Positive responses indicate a positive perception towards injury prevention programs, except the barrier subscale where positive responses indicate a negative perception towards injury prevention programs.
Participant engagement | at 6 weeks
  The participant engagement survey will contain Likert Scale (1-5) questions to provide a quantitative analysis of satisfaction with the program. A 1 indicates strongly disagree and a 5 indicates strongly agree. The range is 7-35, and higher scores indicate increased engagement.
Compliance | 6 weeks
  Compliance will be based on the percentage of sessions attended by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ke'La Porter, MS, ATC,CSCS, Principal Investigator — University of Kentucky
Locations (1):
- Sports Medicine Research Institute, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No